CLINICAL TRIAL: NCT02698059
Title: A Multi-center, Two-stage, Single-arm, Prospective, First-night Order Cross-over, Evaluator-blind Study to Evaluate the Efficacy, Safety and Tolerance of the iNAP® Sleep Therapy System in Adults With Obstructive Sleep Apnea (OSA)
Brief Title: A Post-marketing Surveillance of the Negative Pressure Sleep Therapy System to Treat Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Somnics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: iNAP®-CE-1501
Record Dates: First submitted 2016-02-17; First posted 2016-03-03 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treated (Experimental): iNAP® Sleep Therapy System Treatment
  Interventions: Device: iNAP® Sleep Therapy System (iNAP)
- Baseline/Control (No Intervention): Self-controlled, pre-treatment baseline

INTERVENTIONS:
Device: iNAP® Sleep Therapy System (iNAP) — The iNAP provides pressure gradient within the oral cavity to pull the tongue toward upper palate and the soft palate forward, which aims to maintain better upper airway patency near the pharynx to prevent sleep-disordered breathing.
  Arms: Treated

SUMMARY:
This is a post-marketing surveillance study to investigate the efficacy and safety of the Negative Pressure Sleep Therapy System for the treatment of obstructive sleep apnea.

DETAILED DESCRIPTION:
This is a multi-center, two-stage, single-arm, prospective, first-night order cross-over, evaluator-blind, post-marketing surveillance study to evaluate the efficacy, safety and tolerance of the iNAP® Sleep Therapy System (iNAP), a tongue and soft palate retaining intraoral device, in adults with obstructive sleep apnea (OSA).

ELIGIBILITY:
Inclusion Criteria:

* 1) Female or male adults with age between 18~65 years old. (S1)
* 2) Non-obese patients with body mass index (BMI) <29 kg/m2. (S1)
* 3) Patients able to read and sign on the informed consent form and able to comply with study requirements. (S1)
* 4) Patients able to be properly fitted* with the oral interface as observed by the device feasibility test. (S1)
* 5) Patients with oxygen desaturation index (ODI) between 10~40 (S2).
* 6) Patients with oral negative vacuum time maintained* by iNAP® ≥4 hours/night and total sleep time (TST) ≥4 hours/night (S3).

  * iNAP® pressure more negative than -30 mmHg will be considered evidence of effective oral appliance application.
* 7) Patients with apnea-hypopnea index (AHI) between 10~40 and TST ≥4 hours/night (Baseline PSG Night).
* 8) Patients with oral negative vacuum time maintained* by iNAP® ≥4 hours/night and TST ≥4 hours/night (1st Tx PSG Night).

  * iNAP® pressure more negative than -30 mmHg will be considered evidence of effective oral appliance application.

Exclusion Criteria:

* 1) Patients who are allergic to silicone.
* 2) Patients with obstructed nasal passages as evidenced by the inability to breathe through the nose with the mouth closed.
* 3) Patients who recently experienced a near-miss or prior automobile accident due to sleepiness.
* 4) Patients who have or have had hypoxemia (SpO2 <80%) in the past six months caused by diseases other than OSA such as cardiac disease or severe pulmonary/respiratory disorders such as chronic obstructive pulmonary disease (COPD), interstitial lung disease, pneumothorax, pneumonia, etc.
* 5) Female patients who are lactating, pregnant or intend to become pregnant during the study period.
* 6) Patients with primary insomnia or any concomitant diagnosed or suspected sleep disorder.
* 7) Patients with muscle disease, central nervous disease or chronic neurological disorders, including central sleep apnea*.

  * Central sleep apnea is defined as a central apnea index (CAI) ≥ 5/hr or if central sleep apnea accounts for ≥ 50% of the total AHI.
* 8) Patients in whom it is not suitable to use iNAP® in the opinion of the Investigator including, but not limited to, alcohol or substance abuse, loose teeth, missing teeth, or grinding teeth, completed deviated septum (Type IV or VII) or completed closed nostrils or advanced periodontal disease or tonsillar volumes greater than grade 3.
* 9) Patients with an inability to sleep through the night including, but not limited to, menopausal hot flashes, working at nights or rotating night shifts, planned travel across four or more time zones during the study period or within one week prior to study participation, or a sleep schedule not compatible with study site practices.
* 10) Patients with potential complications of sleep apnea that, in the opinion of the Investigator, may affect the study interpretation or the health or safety of the patients including, but not limited to, narcolepsy, restless leg syndrome, nasopharyngeal carcinoma (NPC), end stage renal failure, a history of severe cardiovascular disease (including New York Heart Association (NYHA) class III or IV cardiac failure, coronary artery disease with angina or myocardial infarction/stroke in the past six months, uncontrolled hypertension or hypotension or cardiac arrhythmias), unstable heart or renal transplantation or use of medicine or other treatment(s) that may confound the result of the study or pose additional risks to the patient, such as oral anticoagulants or other agents making patients prone to tongue hemorrhage.

Stage II Inclusion Criteria:

Patients who fulfill all the enrollment criteria of Stage I and whose treated AHI on the 1st Tx PSG Night is below 40.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2016-01-22 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate* of apnea-hypopnea index (AHI)** on the 1st Tx PSG Night when compared to the Baseline PSG Night. | first treatment night
  *Clinical success rate is defined as the ratio of the number of patients with an AHI reduction of >50% and treated AHI <20 to the number of patients who complete the 1st Tx PSG Night, where completion is defined as a total sleep time (TST) and device negative pressure maintenance ≥4 hours/night on the 1st Tx PSG Night. For completion of the Baseline PSG Study, a total sleep time (TST) ≥4 hours/night has to be met.
  **AHI is the number of apnea/hypopnea events divided by total sleep time (TST), i.e., the number of hours of sleep.

SECONDARY OUTCOMES:
AE/SAE rate and type | The whole study period through study completion; up to 8 weeks
  Vital signs, Physical examination (PE) findings and change of body figure indexes, Electrocardiogram (ECG) findings as reflected in polysomnography (PSG), Adverse events (AEs), Serious adverse events (SAEs), Changes in the oral and dental condition
Clinical success rate* of apnea-hypopnea index (AHI)** on the 2nd Tx PSG Night when compared to the 1st Tx PSG Night. | second treatment night
  *Clinical success rate is defined as the ratio of the number of patients with an AHI reduction of >50% and treated AHI <20 to the number of patients who complete the 2nd Tx PSG Night, where completion is defined as a total sleep time (TST) and device negative pressure maintenance ≥4 hours/night on the 2nd Tx PSG Night. For completion of the Baseline PSG Study, a total sleep time (TST) ≥4 hours/night has to be met.
  **AHI is the number of apnea/hypopnea events divided by total sleep time (TST), i.e., the number of hours of sleep.
Change of Oxygen Desaturation Index (ODI)* from the Baseline PSG Night compared to the 1st Tx PSG Night and the 2nd Tx PSG Night; and the change from the 1st Tx PSG Night compared to the 2nd Tx PSG Night. | At the Baseline PSG Night, the 1st Tx PSG Night and/or the 2nd Tx PSG Night
  *ODI is the event number of oxygen level drops by 3 percent or more from baseline divided by total sleep time (TST), i.e., the number of hours of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Schneider, M.D., Principal Investigator — American Sleep Clinic Frankfurt
Locations (8):
- Germany (6):
  - INTERSOM, Cologne
  - Somnolab, Dortmund
  - Alfred Krupp Krankenhaus, Essen
  - American Sleep Clinic, Frankfurt
  - HELIOS Klinik Ambrock, Hagen
  - Krankenhaus Bethanien, Solingen
- Taiwan (2):
  - Mackay Memorial Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilius G, Farid-Moayer M, Lin CM, Knaack L, Wang YP, Dellweg D, Stoohs R, Ficker J, Randerath W, Specht MB, Galetke W, Schneider H; iNAP Study Group. Multi-center safety and efficacy study of a negative-pressure intraoral device in obstructive sleep apnea. Sleep Med. 2024 Jul;119:139-146. doi: 10.1016/j.sleep.2024.04.015. Epub 2024 Apr 17. PMID 38678757